CLINICAL TRIAL: NCT01284140
Title: Improving the Sleep and Circadian Rhythms of Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian Gehlbach (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Brian Gehlbach, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201105754; 5K23HL088020 (NIH)
Record Dates: First submitted 2011-01-19; First posted 2011-01-26 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Critical Illness; Sleep Deprivation; Respiratory Failure; Sleep Disorders, Circadian Rhythm
Keywords: Critical illness; Sleep; Polysomnography; Respiratory failure; Circadian rhythm; Sedation
MeSH Terms: conditions — Critical Illness; Sleep Deprivation; Respiratory Insufficiency; Sleep Disorders, Circadian Rhythm | interventions — Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleep promotion protocol (Experimental): Behavioral: 48 hours of sleep and circadian rhythm promotion including timed light exposure.
  Interventions: Behavioral: Sleep and circadian rhythm promotion
- Usual care (Active Comparator): Behavioral: 48 hours of usual care.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Sleep and circadian rhythm promotion — This multifaceted intervention attempts to enhance sleep and circadian rhythmicity through improved scheduling of nursing procedures, enforcement of a day/night routine, increased light exposure during the day, and decreased light and sound exposure during the night. The intervention began the morning after enrollment and enforced a specific period of enhanced light exposure from 9:00 a.m. to noon. The initial target of 5,000 lux administered by light box (Sunsation, SunBox Co.) was reduced to 400-700 lux after the first 10 subjects were enrolled in the study.
  Arms: Sleep promotion protocol
Behavioral: Usual care — Usual care.
  Arms: Usual care

SUMMARY:
The goal of this project is to determine whether the sleep and circadian rhythms of critically ill patients undergoing mechanical ventilation can be improved through practical strategies that can be employed at the bedside.

DETAILED DESCRIPTION:
Nearly 1 million patients develop respiratory failure annually in the United States; yet, the sleep of patients undergoing mechanical ventilation has received little attention. This project is designed to characterize sleep and circadian rhythmicity in critically ill patients and to explore the efficacy of a non-pharmacological intervention to improve sleep and normalize circadian phase. The study will examine the effect of a protocol employing noise reduction and enforcement of a robust light-dark cycle on sleep quality and circadian rhythmicity. A secondary analysis will examine the relationship between delirium and sleep disruption and loss of circadian rhythmicity. Circadian rhythmicity will be characterized through the measurement of urinary 6-sulfatoxymelatonin levels at frequent intervals, while sleep will be assessed using continuous polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Receiving mechanical ventilation and intravenous sedation

Exclusion Criteria:

* Debilitating central nervous system disease or degenerative disorder
* Active seizures
* Persistent coma
* Renal failure requiring dialysis
* Expected to be extubated within 24 hours
* Currently receiving neuromuscular blocker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian K Gehlbach, MD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the medical intensive care units of the University of Chicago and the University of Iowa Hospitals and Clinics.
Pre-assignment Details: Two subjects who acutely developed exclusion criteria were withdrawn from the study after enrollment and prior to the performance of any study-related procedures. These subjects were not analyzed.
Period: Randomization and Intervention
Arm/Group | Sleep Promotion Protocol | Usual Care
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Subjects With Paired 24hr Collections
Arm/Group | Sleep Promotion Protocol | Usual Care
Started | 11 | 11
Completed | 6 | 5
Not Completed | 5 | 6
Not completed — Day 3 urinary profile not available | 5 | 5
Not completed — Day 1 urinary profile incomplete | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects with 24-hour urinary 6-sulfatoxymelatonin profiles from both Day 1 and Day 3 were analyzed (11 subjects out of a total of 22). One of the remaining subjects had an unevaluable profile from Day 1. The remaining subjects died or had their urinary catheter removed prior to Day 3.
Groups:
- Sleep Promotion Protocol: Behavioral: sleep and circadian rhythm promotion including timed light exposure.
  Sleep and circadian rhythm promotion: This multifaceted intervention will attempt to enhance sleep and circadian rhythmicity through improved scheduling of nursing procedures, enforcement of a day/night routine, increased light exposure during the day, and decreased light and sound exposure during the night. Supplemental bright lights and eyeshades and noise cancelling headphones may also be employed.
- Usual Care: Behavioral: usual care.
  Usual care: Usual care.
- Total: Total of all reporting groups
Arm/Group | Sleep Promotion Protocol | Usual Care | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (10.4) | 59.6 (7.7) | 63.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Acute Physiology and Chronic Health Evaluation II score [Mean (Standard Deviation); unit: units on a scale] — The Acute Physiology and Chronic Health Evaluation (APACHE) II score is a severity of illness score that estimates ICU mortality. An integer score from 0 to 71 is computed based on several measurements, with higher scores corresponding to higher predicted mortality.
  units on a scale | 25.5 (2.5) | 24.4 (2.0) | 25 (5.3)
Mechanically ventilated during study period [Count of Participants; unit: Participants] | 6 | 5 | 11
Total urinary 6-sulfatoxymelatonin excretion on day 1 (micrograms) [Mean (Standard Deviation); unit: micrograms] | 14.5 (4.7) | 20.4 (8.1) | 17.2 (14.5)
Body mass index [Median (Inter-Quartile Range); unit: kg per meters squared] | 25.0 [21.8 to 33.2] | 27.4 [26.0 to 37.9] | 26.4 [24 to 35.5]
Average peak creatinine during study period [Mean (Standard Deviation); unit: mg per deciliter] | 2.0 (0.6) | 1.8 (0.5) | 1.9 (1.3)
Propofol during study period [Count of Participants; unit: Participants] | 6 | 5 | 11
Opioids during study period [Count of Participants; unit: Participants] | 6 | 5 | 11
Benzodiazepines during study period [Count of Participants; unit: Participants] | 0 | 3 | 3
Dexmedetomidine during study period [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Circadian Timing
Description: The magnitude of the phase change in 6-sulfatoxymelatonin excretion between Day 1 and Day 3 will be compared between the intervention and usual care groups. This is done by comparing, for each group, the timing of the best-fit maximum on Day 1 with the timing of the best-fit maximum on Day 3. The result is expressed in hours. A positive value represents a phase advance from Day 1 to Day 3 (e.g. an earlier occurrence of maximum excretion on Day 3 when compared with Day 1), while a negative value represents a phase delay from Day 1 to Day 3 (e.g. a later occurrence of maximum excretion on Day 3 when compared with Day 1).
Time Frame: Day 1 to Day 3
Population: Subjects with 24-hour 6-sulfatoxymelatonin excretion profiles from both Day 1 and Day 3.
Measure: Number; unit: hours
Arm/Group | Sleep Promotion Protocol | Usual Care
Number analyzed (Participants) | 6 | 5
hours | 3.6 | -2.4
Statistical Analysis 1: Comparison: Usual Care; Nonlinear regression using the least-squares approach was used to fit a single 24-hour cosine curve to all normalized data in each group on each day of 24-hour urine collection. Model parameters of acrophase and amplitude and their standard errors were derived from these curves. Using the extra sum-of-squares F test, the null hypothesis that model parameters of amplitude and phase were the same on Day 1 and Day 3 was tested for the Usual Care group; Test type: Other; p = 0.37, Extra sum-of-squares F test; The null hypothesis that model parameters of amplitude and phase were the same on Day 1 and Day 3 was not rejected for the Usual Care group
Statistical Analysis 2: Comparison: Sleep Promotion Protocol; Nonlinear regression using the least-squares approach was used to fit a single 24-hour cosine curve to all normalized data in each group on each day of 24-hour urine collection. Model parameters of acrophase and amplitude and their standard errors were derived from these curves. Using the extra sum-of-squares F test, the null hypothesis that model parameters of amplitude and phase were the same on Day 1 and Day 3 was tested for the Sleep promotion group; Test type: Other; p = 0.0074, Extra sum-of-squares F test; This result suggests that the best-fit values for amplitude and phase are different between Day 1 and Day 3 in the Sleep Promotion group

2. Secondary Outcome: Normal Circadian Timing
Description: The percentage of subjects who exhibit normal circadian timing of 6-sulfatoxymelatonin excretion on Day 3 will be compared between the intervention and usual care groups.
Time Frame: Day 3
Population: Subjects with 24-hour 6-sulfatoxymelatonin excretion profiles from both Day 1 and Day 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Promotion Protocol | Usual Care
Number analyzed (Participants) | 6 | 5
Participants | 3 | 1
Statistical Analysis 1: Comparison: Sleep Promotion Protocol vs Usual Care; Test type: Superiority; p = 0.55, Fisher Exact

3. Secondary Outcome: Circadian Amplitude
Description: The amplitude (e.g. one half the value from peak to trough of the fitted cosine curve) of the circadian rhythm of 6-sulfatoxymelatonin on Day 3 will be compared between the usual care and intervention groups.
Time Frame: Day 3
Population: Subjects with 24-hour 6-sulfatoxymelatonin excretion profiles from both Day 1 and Day 3.
Measure: Mean (Standard Deviation); unit: percent of 24-hour mean 6-sulfatoxymelat
Arm/Group | Sleep Promotion Protocol | Usual Care
Number analyzed (Participants) | 6 | 5
percent of 24-hour mean 6-sulfatoxymelat | 36.6 (14.5) | 11.0 (17.7)
Statistical Analysis 1: Comparison: Sleep Promotion Protocol vs Usual Care; Nonlinear regression using the least-squares approach was used to fit a single 24-hour cosine curve to all normalized data in each group on each day of 24-hour urine collection. This resulted in 4 separate best-fit curves. The model parameter of amplitude was derived from the best-fit curves; Test type: Superiority; p = 0.03, t-test, 2 sided; Mean Difference (Final Values) = 0.03

4. Secondary Outcome: Spectral Edge Frequency 95%
Description: The difference between the polysomnographically derived daytime and nocturnal spectral edge frequency 95% parameter will be used as a measure of increased diurnal sleep/wake activity. This parameter will be compared between the usual care and intervention groups.
Time Frame: Day 2
Population: Polysomnography was not conducted on any participants due to logistical constraints.
Arm/Group | Sleep Promotion Protocol | Usual Care
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Delirium
Description: The percentage of patients who are delirious at the conclusion at the study will be compared between the intervention and usual care groups.
Time Frame: Day 3
Population: Subjects still on study in the ICU on Day 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Promotion Protocol | Usual Care
Number analyzed (Participants) | 6 | 5
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: From the day of enrollment until the completion of all bedside assessments 3 days later.
Arm/Group | Sleep Promotion Protocol | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/11 | 2/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Lower dose light intervention received by one subject; the study design resulted in significant attrition, limiting the number of evaluable patients; baseline differences in the timing of maximal melatonin excretion may have influenced the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No